CLINICAL TRIAL: NCT06211140
Title: Effect of Transcranial Alternating Current Stimulation (tACS) on Serotonin-1A Receptor in Patients With Major Depressive Disorder
Brief Title: Transcranial Alternating Current Stimulation (tACS) on Serotonin-1A Receptor in Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tACS-MDD
Record Dates: First submitted 2023-12-19; First posted 2024-01-18 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; tACS; 5-HT
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; Non-Randomized; Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depressive disorders (Experimental): Three conductive electrodes will be placed overhead. Based on the 10/20 international placement system, a 4.45 x 9.53 cm electrode is placed on the forehead corresponding to Fpz, Fp1 and Fp2. Two 3.18 x 3.81 cm electrodes are placed on the mastoid region of each side.
  The tACS stimulation waveform includes ramp-up and ramp-down periods of 180 and 12 s, respectively. It is a square-wave with an average amplitude of 15 mA and is equally distributed from the frontal region to the mastoid areas (amplitudes are reported as zero-to-peak).
  All participants with major depression disorder will receive a total of 20 sessions in four weeks, once daily on weekdays, with tACS stimulation at 77.5 Hz and 15 mA.
  From Monday to Friday, each session will last 40 min at a fixed daytime interval.
  Interventions: Device: tACS
- Healthy controls (Other): Without the tACS stimulation in this group
  Interventions: Other: Control

INTERVENTIONS:
Device: tACS — tACS in 4 weeks, once per weekday for 40 minutes each, 20 sessions. The treatment group will receive transcranial alternating current stimulation at a gamma frequency (77.5Hz) with a peak amplitude of 15mA.
  Arms: Depressive disorders
Other: Control — Without the tACS stimulation in this group.
  Arms: Healthy controls

SUMMARY:
This study will apply a comprehensive tools that integrates neuroimaging, psychological evaluation, and sleep monitoring through 18F-MPPF PET/MR, neuropsychological tests, and polysomnography (PSG) to explore the neurobiological mechanisms underlying transcranial alternating current stimulation (tACS) for depressive disorders, mainly focusing on the serotonergic system revealed by Serotonin-1A (5-HT1A) receptor.

DETAILED DESCRIPTION:
5-HT1A receptor appears to be significantly involved in the effectiveness of electroconvulsive therapy (ECT). Like alternating current in ECT, tACS also applies alternating current to intervene in neuropsychiatric disorders. We previously found that tACS with large current, such as 15 mA, via the forehead and bilateral mastoids can improve depressive symptoms. However, the underlying mechanism of 15 mA tACS in depression remains unclear. We propose a scientific hypothesis that 15 mA tACS may increase hippocampal 5- HT1A receptors, then to reduce depression in depressive patients. Meanwhile, 15 mA tACS may increase the whole-brain functional connectivity with the hippocampus as the seed point. This study will utilize a multimodal data through 18F-MPPF PET/MR, including MPPF metabolism, resting-state fMRI, DTI, and 3D-T1 structural images. By observing the alterations of 5-HT1A receptor and the functional network between MDD patients and healthy controls, and between the pre- and post-tACS intervention in MDD patients, our aims to explore the effect of tACS on the serotonergic system in depression.

ELIGIBILITY:
Inclusive Criteria:

1. 18 to 65 years old, Chinese, male or female.
2. Non-psychotic major depressive disorder according to DSM-IV.
3. HAMD-17 total score ≥ 17 at the baseline.
4. Currently experiencing an acute episode.
5. No history of prior treatment with psychotropic medications.
6. Understanding of all aspects of the research protocol and the ability to provide informed consent.

Exclusion Criteria for patients:

1. Unable to do PET/MR examinations.
2. Have secondary insomnia disorders, anxiety disorders, or depressive disorders caused by physical illnesses.
3. Severe or unstable organic diseases.
4. Pregnant or lactating women or those planning a pregnancy in the near future.
5. Alcohol or substance dependence or abuse within the past year.
6. Received electroconvulsive therapy or transcranial magnetic stimulation in the month preceding enrollment.
7. Skin damage at the electrode placement site or those allergic to electrode gel or adhesives.
8. Participated in any other clinical trials within the month before baseline.
9. Any inappropriate conditions considered by the study group.

Inclusion Criteria for healthy volunteers

1. To undergo PET/MR examinations.
2. Be matched with the patient group regarding age, sex, and educational level.

Exclusion Criteria for healthy volunteers:

1. Those who are enrolled in other clinical studies.
2. The inappropriate conditions considered by the study group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The changes in quantitative MPPF values before and after the tACS intervention. | baseline (before the tACS intervention), 4 weeks (after the tACS intervention)
  Twenty patients with depressive disorders will receive 18F-MPPF PET/MR imaging before and after the tACS intervention. MPPF metabolism values in different brain regions will be calculated.
  A comparative analysis will be then performed between the baseline and post-treatment in patients with depressive disorders.

SECONDARY OUTCOMES:
The changes in scores for 17-item Hamilton Depression Rating Scale (HAMD-17) before and after the tACS intervention. | baseline, 4 weeks
  HAMD-17 will be assessed before and after the tACS intervention in twenty patients with depressive disorders. HAMD-17 scores range from 0 to 52, with higher scores indicating more depression, a score of 24 or more indicates severe depression.
The changes in scores for Hamilton Anxiety Rating Scale (HAMA) before and after the tACS intervention. | baseline, 4 weeks
  HAMA evaluation will be conducted before and after the tACS intervention in twenty patients with depressive disorders. HAMA scores range from 0 to 56, with higher scores indicating more anxiety, a score of 29 or more indicates severe anxiety.
The changes in scores for Generalized Anxiety Disorder-7 item (GAD-7) before and after the tACS intervention. | baseline, 4 weeks
  GAD-7 total score range 0 to 21. A score of 10 or higher means significant anxiety is present. Score over 15 are severe.
The changes in scores for Pittsburgh Sleep Quality Index (PSQI) before and after the tACS intervention. | baseline, 4 weeks
  PSQI score ranges 0 to 21, a score of 8 or more indicates insomnia.
The changes in scores for Insomnia Severity Index (ISI) before and after the tACS intervention. | baseline, 4 weeks
  ISI total score is 0 to 28, a total score of 0-7 indicates 'no clinically signifi cant insomnia', 8-14 means 'subthreshold insomnia', 15-21 is 'clinical insomnia (moderate severity)', and 22-28 means 'clinical insomnia (severe)'.
Cognitive changes will be assessed using the Montreal Cognitive Assessment (MoCA) before and after the tACS intervention in depression. | baseline, 4 weeks
  MoCA total score ranges 0 to 30. If the length of education is less than 12 years, 1 point will be added, with a maximum score of 30 points. A score of 26 is considered normal.
Cognitive changes will be assessed using the Mini-Mental State Examination (MMSE) before and after the tACS intervention in depression. | baseline, 4 weeks
  MMSE total score is from 0 to 30. The criteria on cognitive impairment in Chinese as follows: the illiterate ≤ 17 points, the primary school ≤ 20 points, and the middle school or above ≤ 24 points

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China